CLINICAL TRIAL: NCT05918341
Title: The Feasibility of Using a Subtherapeutic Dose of Piracetam as a Marker of Adherence to Therapy
Brief Title: Subtherapeutic Dose of Piracetam as a Therapy Adherence Marker
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N23PIR
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Drug Adherence Marker
Keywords: Drug adherence, adherence tracer, subtherapeutic dosing, quantitative urinalysis
MeSH Terms: conditions — Medication Adherence | interventions — Piracetam

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open-label, uncontrolled study in 10 healthy volunteers who will receive various subtherapeutic doses of piracetam.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Piracetam arm (single arm) (Experimental): The single to take once weekly doses of 7.5 mg, 5 mg, 2.5 mg and 1.25 mg piracetam consecutively. Urine was collected 24 and 72 hours after the weekly doses were taken. It was chosen to administer all these doses in each healthy volunteer to account for inter-individual differences in urine concentrations, as these concentrations depend on individual characteristics such as volume intake and renal function.
  Interventions: Drug: Piracetam

INTERVENTIONS:
Drug: Piracetam — Subtherapeutic dose of piracetam (once-weekly doses of 7.5 mg, 5 mg, 2.5 mg and 1.25 mg)

SUMMARY:
The aim of this study is to test a subtherapeutic dose of piracetam in healthy volunteers as a marker of adherence to therapy to assess the feasibility of its use in a multicentre, randomised, double-blind, placebo-controlled study of the efficacy of dexamphetamine in cocaine dependence (CUD) with comorbid opioid addiction (REDUCE study). Several markers for assessing adherence have been described in the literature. However, none of these markers qualified for use within the targeted patient population. Therefore, a suitable adherence marker was sought specifically for the study design of the REDUCE trial. Since within the REDUCE trial urine is submitted biweekly by participants for measuring cocaine use, the adherence marker will also be determined in this matrix. The most suitable marker seems to be piracetam. However, within this study with healthy volunteers, it will first have to be confirmed whether detectable concentrations of piracetam are actually excreted in the urine.

DETAILED DESCRIPTION:
This study with healthy volunteers will test a subtherapeutic dose of piracetam as an adherence marker to assess the feasibility of its use in a multicenter, randomized, double-blind, placebo-controlled study of the efficacy of dexamfetamine in cocaine use disorder (CUD) with comorbid opioid use disorder (REDUCE-trial).

Adherence to the study medication in the REDUCE-trial will be assessed by urinanalysis twice weekly for the presence of dexamfetamine. To determine adherence in the placebo group, the tablets must be formulated with a marker detectable in urine. It is necessary to assess adherence in the clinical trial since stimulants will be provided to patients who are dependent on stimulants. Moreover, monitoring adherence ensures that efficacy is established when the medication is taken at the correct dose and frequency.[1] Non-adherence to study medication is especially a problem in trials involving the addicted population, with 10% of participants never taking a dose.[2] In addition, relatively low adherence rates (39-42%) are common for this population.[3][4] Efficacy and safety effects may be underestimated as a result of nonadherence to study medication. Since adherence to placebo was found to be a predictor of better treatment outcomes, it is important to assess this as well.[5]

Several markers for assessing medication adherence are described in the literature.[1][7-12] However, none of these previously used markers were eligible for use within the clinical trial design. First, the measurement of adherence for some markers was based on urine staining (methylene blue, phenol red, fluorescein, phenazopyridine) that would be visible to patients enrolled in the trial. Second, some markers (riboflavin, quinine) are interfered with by dietaryor vitamin intake.[1] In addition, some markers are limited by the occurrence of side effects (phenobarbital).[10][11] Finally, the long half-life of the adherence markers bromide and digoxin would not fit the twice weekly urinalysis, where non-compliance of several days would be masked.[7-9] Therefore, a suitable marker for the clinical trial was searched.

The ideal marker is nontoxic and potentially detectable in urine at a subtherapeutic dose. Therefore, a drug with a relatively high therapeutic dose, high bioavailability, high unchanged renal clearance and low hepatic metabolism is favourable. Thus, detectable amounts in urine at subtherapeutic dose would be likely. Moreover, the half-live of the marker must match the twice weekly assessments of adherence. Of all the authorised drugs in the Netherlands, piracetam was found to meet the most of the criteria. Piracetam is a well-tolerated therapy and registered in the Netherlands for the treatment of vertigo. Daily therapeutic intake is 2400 mg with complete bioavailability, no hepatic metabolism and a renal clearance of about 90%.[13] The likelihood of interference with prescribed piracetam is low, as only 740 patients used the drug in the Netherlands in 2021.[14]

The subtherapeutic dose of piracetam was calculated using the EMA guidelines on shared manufacturing facilities.[15] This guideline contains acceptance limits of cross-contamination between drugs in multipurpose manufacturing processes. These limits are based on the absence of a therapeutic or toxicological effect of the residues of an active drug.[15] The permitted daily exposure (PDE) is calculated using all available pharmacological and toxicological data, including both non-clinical and clinical data, to derive safe thresholds. The PDE represents a substance-specific dose that is unlikely to cause adverse effects if a person is exposed to or below this dose for a lifetime. The PDE for piracetam was calculated to be 8 mg (Appendix I). As patients in the clinical trial receive one, two or three placebo tablets per day, the intention is to add 2.5 mg of piracetam to the placebo tablets. If the urine concentration of piracetam known in the literature at daily intake of 800 mg is extrapolated to 2.5 mg, a measurable urine concentration of 200 ng/ml is expected.[16] However, it should first be confirmed in healthy volunteers whether detectable piracetam concentrations are actually excreted in the urine.

References

1. Babalonis S, Hampson AJ, Lofwall MR, Nuzzo PA, Walsh SL. Quinine as a potential tracer for medication adherence: A pharmacokinetic and pharmacodynamic assessment of quinine alone and in combination with oxycodone in humans. J Clin Pharmacol. 2015 Dec;55(12):1332-43. doi: 10.1002/jcph.557. Epub 2015 Jul 29. PMID: 26032168; PMCID: PMC4666817.
2. Anderson AL, Li SH, Biswas K, et al. Modafinil for the treatment of methamphetamine dependence. Drug Alcohol Depend. 2012; 120(1-3):135-141. [PubMed: 21840138]
3. Swift R, Oslin DW, Alexander M, Forman R. Adherence monitoring in naltrexone pharmacotherapy trials: a systematic review. J Stud Alcohol Drugs. 2011; 72(6):1012-1018. [PubMed: 22051215]
4. Weiss RD. Adherence to pharmacotherapy in patients with alcohol and opioid dependence. Addiction. 2004; 99(11):1382-1392. [PubMed: 15500591]
5. Granger BB, Swedberg K, Ekman I, et al. Adherence to candesartan and placebo and outcomes in chronic heart failure in the CHAEM prgramme: double-blind, randomized, controlled clinical trial. Lancet. 2005; 366(9502):2005-11. [PubMed: 16338449]
6. Ritscher S, Georges C, Wunder C, Wallemacq P, Persu A, Toennes SW. Assessment of adherence to diuretics and β-blockers by serum drug monitoring in comparison to urine analysis. Blood Press. 2020 Oct;29(5):291-298. doi: 10.1080/08037051.2020.1763775. Epub 2020 May 13. PMID: 32400211.
7. Braam RL, van Uum SH, Lenders JW, Thien T. Bromide as marker for drug adherence in hypertensive patients. Br J Clin Pharmacol. 2008 May;65(5):733-6. doi: 10.1111/j.1365-2125.2007.03068.x. Epub 2008 Feb 12. PMID: 18279473; PMCID: PMC2432484.
8. Braam RL, van Uum SH, Russel FG, Swinkels DW, Thien T. Bromide as a marker to measure adherence to drug therapy. Eur J Clin Pharmacol. 2006 Apr;62(4):285-90. doi: 10.1007/s00228-006-0103-5. Epub 2006 Mar 7. PMID: 16525815.
9. Mäenpää H, Javela K, Pikkarainen J, Mälkönen M, Heinonen OP, Manninen V. Minimal doses of digoxin: a new marker for compliance to medication. Eur Heart J. 1987 Oct;8 Suppl I:31-7. doi: 10.1093/eurheartj/8.suppl_i.31. PMID: 3322828.
10. Feely M, Cooke J, Price D, Singleton S, Mehta A, Bradford L, Calvert R. Low-dose phenobarbitone as an indicator of compliance with drug therapy. Br J Clin Pharmacol. 1987 Jul;24(1):77-83. doi: 10.1111/j.1365-2125.1987.tb03139.x. PMID: 3113467; PMCID: PMC1386283.
11. Wolff K, Hay AA, Raistrick D, Feely M. Use of 'very low-dose phenobarbital' to investigate compliance in patients on reducing doses of methadone (detoxification). J Subst Abuse Treat. 1993 SepOct;10(5):453-8. doi: 10.1016/0740-5472(93)90006-n. PMID: 8246320.
12. Herron AJ, Mariani JJ, Pavlicova M, Parrinello CM, Bold KW, Levin FR, Nunes EV, Sullivan MA, Raby WN, Bisaga A. Assessment of riboflavin as a tracer substance: comparison of a qualitative to a quantitative method of riboflavin measurement. Drug Alcohol Depend. 2013 Feb 1;128(1-2):77-82. doi: 10.1016/j.drugalcdep.2012.08.007. Epub 2012 Aug 22. PMID: 22921475; PMCID: PMC3556739.
13. KNMP Kennisbank. (2022). Informatorium Medicamentorum (Piracetam). Accessed on 21th of December 2022
14. Zorginstituut Nederland (ZIN). GIP databank. 2023. Available: Aantal gebruikers 2017-2021 voor ATC-subgroep N06BX03 : Piracetam | GIPdatabank.nl [Accessed 23 March 2023]
15. European Medicine Agency (EMA). EU GMP guide part I: basic requirements for medicinal products: Chapter 3: Shared Manufacturing facilities. 2015. Available: Guideline on setting health based exposure limits for use in risk identification in the manufacture of different medicinal products in shared facilities (europa.eu) [Accessed 23 March 2023]
16. Louchahi K, Tod M, Bonnardel P, Petitjean O. Determination of piracetam in human plasma and urine by liquid chromatography. J Chromatogr B Biomed Appl. 1995 Jan 20;663(2):385-9. doi: 10.1016/0378-4347(94)00448-e. PMID: 7735487.
17. College ter Beoordeling Geneesmiddelen (CBG). Geneesmiddeleninformatiebank. 2023. Available: https://www.geneesmiddeleninformatiebank.nl/smpc/h18655_smpc.pdf [Accessed 23 March 2023]

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Able and willing to give written informed consent;
3. Able and willing to undergo urine sampling for analysis;
4. Able and willing to digest multiple tablets at day one of each study week (6 tablets of 1.25 mg in week 1; 4 tablets of 1.25 mg in week 2; 2 tablets of 1.25 mg in week 3 and 1 tablet of 1.25 mg in week 4.

Exclusion Criteria:

1. Current prescribed treatment with piracetam;
2. Pregnant or breastfeeding;
3. Criteria regarding the following contra-indications for piracetam:

   * Cerebral haemorrhage;
   * Huntington's chorea;
   * Hypersensitivity to pyrrolide derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-03 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective (detectability of piracetam in urine) | 24 hours after weekly ingestion of weekly dosage
  To assess the feasibility of using a subtherapeutic dose of piracetam as a marker of adherence to therapy by determining whether this subtherapeutic dose produces a detectable concentration in the urine.

SECONDARY OUTCOMES:
Secondary Objective (piracetam concentration after nonadherence) | 72 hours after weekly ingestion of weekly dosage
  To determine the piracetam urine concentrations after nonadherence of two days.

CONTACTS AND LOCATIONS:
Overall Officials: Alwin Huitema, Prof. Dr., Principal Investigator — The Netherlands Cancer Institute

IPD SHARING:
Plan to Share IPD: No
Providing raw participant data to other researchers, for this particular study, will not be of general interest. However, all measured urine concentrations will be published and can be accessed by other researchers in this way.